CLINICAL TRIAL: NCT06902142
Title: Étude Multicentrique Prospective de la Relation Entre Efficacité Virologique et Observance Chez Des Patients Infectés Par le VIH-1 Traités Par Bictegravir
Brief Title: Prospective Multicenter Study of the Relationship Between Virological Effectiveness and Compliance in HIV-1-infected Patients Treated With Bictegravir
Acronym: BICTECAPS
Status: Recruiting | Type: Observational
Sponsor: Association pour la promotion de la recherche en maladies infectieuses et tropicales dans le Loiret (Other)
Collaborators: Hôpital Côte de Nacre, CHU de Caen (Unknown)
Responsible Party: Principal Investigator, Laurent HOCQUELOUX, MD, Investigator coordinator, Centre Hospitalier Régional d'Orléans
Other Study IDs: APREMIT 45 (04); CO-FR-380-7223 (Other Grant/Funding Number: GILEAD SCIENCES); 2024-A01111-46 (Other: ID RCB)
Record Dates: First submitted 2025-03-14; First posted 2025-03-30 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-02

CONDITIONS: HIV Antiretroviral Therapy (ART) Adherence
Keywords: HIV-1; B/F/TAF; Adherence; Forgiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults living with HIV-1 receiving or starting once-daily B/F/TAF-based antiretroviral therapy: Given our interest in covering a wide range of adherence profiles of B/F/TAF, the participation of PLHIV perceived by their physicians to be at risk of suboptimal adherence, such as a history of pre-existing resistance that does not affect B/F/TAF, immigrants/migrants, homeless/poorly housed, those with substance use disorders, transgender women, youth and those facing mental health issues, will be encouraged
  Interventions: Device: Adherence measured by MEMS caps

INTERVENTIONS:
Device: Adherence measured by MEMS caps — The methodological choices made in this study are justified by the need to assess the effectiveness of bictegravir, taking into account the varying levels of adherence among PLHIV. The use of electronic antiretroviral caps (MEMS caps: https://aardexgroup.com/medication-event-monitoring-system/ ) and the intra-cellular TAF assay to measure drug concentrations will enable a combined, precise and objective assessment of treatment adherence, and constitute the originality of this research.

SUMMARY:
Modern once-daily antiretroviral therapies have evolved considerably, improving patients' quality of life. However, sub-optimal adherence to antiretroviral therapy (ART) can lead to insufficient viral suppression and the emergence of resistant HIV strains. In particular, several populations encountered in HIV clinical practice face obstacles to optimal adherence.

The investigators propose the prospective multicenter cohort study BICTECAPS, evaluating the effectiveness of the combination therapy bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) in routine practice. The investigators hypothesize that the pharmacokinetic profile and genetic barrier provided by B/F/TAF will enable a high rate of virological suppression at low to moderate levels of adherence, probably 100% virological suppression above 70% adherence.

The study is planned to include 120 patients with HIV infection treated with B/F/TAF, over a planned 2-year period with usual follow-up.

The aim of this work is to evaluate virological suppression rates at 6 and 12 months according to adherence levels defined by electronic antiretroviral monitoring caps (MEMS caps) and by intra-cellular TAF assay on blotting paper (dried blood spot, DBS).

The investigators hope to generate real-life data on B/F/TAF use from population groups generally under-represented in clinical trials, including robust measurements of adherence patterns using MEMS caps and DBS.

. Key words : HIV-1 ; B/F/TAF ; Adherence ; Forgiveness

DETAILED DESCRIPTION:
Title Etude multicentrique prospective de la relation entre efficacité virologique et observance chez des patients infectés par le VIH-1 traités par BICTEGRAVIR

Type or research Non interventional research (NIR)

Target population People living with HIV (PLWH)

Objectives Primary objective:

- To explore the effectiveness of antiretroviral treatment with B/F/TAF by virological suppression rate (plasma HIV-RNA) at 6 months in real life according to adherence patterns defined by electronic antiretroviral monitoring caps (MEMS caps) and by intra-cellular TAF assay.

Secondary objective(s):

* To explore the effectiveness of antiretroviral treatment with B/F/TAF by the rate of virological suppression (plasma HIV-RNA) at 12 months in real life, according to adherence patterns defined by electronic antiretroviral monitoring caps (MEMS caps).
* Evaluate the risk of emergence of resistance mutations in cases of HIV RNA replication with B/F/TAF.
* Evaluate the safety profile of B/F/TAF in real-life practice.
* Evaluate the quality of life of participants treated with B/F/TAF in real-life practice.

Inclusion Criteria -

* Person living with HIV-1
* 18 years of age or older
* Having been informed about the study (non-opposition)
* Accepts the use of electronic antiretroviral monitoring caps (MEMS caps)
* Person treated or starting treatment with bictegravir/emtricitabine/tenofovir (B/F/TAF; antiretroviral treatment naïve, changing treatment, virological failure) Exclusion criteria -
* Pregnant women
* People living with HIV (PLHIV) unable to assume responsibility for treatment compliance (impaired judgment, guardianship, institutionalization)
* PLWH receiving assistance incompatible with the use of the electronic pillbox

Endpoints

Primary :

- Virological failure at 6 months defined as a confirmed plasma viral load >50 copies/mL or a single plasma viral load >200 copies/mL (HIV RNA).

Secondary :

* Virological failure at 12 months as defined above
* Rate of side effects measured by CTCAE V.5
* Emergence of drug resistance mutations according to ANRS AC11 V35 in case of virological replication
* Quality of life measured by questionnaires

Procedure(s) or visit(s) added by research none

Nomber of patients 120 patients : Accuracy of at least +/-7% on virological failure rate

Number of centers 8 centers :

* CHU CAEN NORMANDIE
* CHU d'Orléans
* APHP Pitié-Salpêtrière
* CHU Poitiers
* CHU Nantes
* CHD La Roche sur Yon
* CH de Niort
* HCL Lyon

Project Milestone

* Expected start date of inclusions: 01/09/2024
* Inclusion duration: 2 years
* Duration of follow-up period: 12 months
* Planned end of study (issue of final report summary 1 year after last visit to last included subject): 01/09/2027

ELIGIBILITY:
Inclusion Criteria:

* People living with HIV-1
* Age greater than or equal to 18 years
* Having been informed about the study (non-opposition)
* Acceptance of the use of electronic antiretroviral monitoring caps (MEMS caps)
* People treated or starting treatment with bictegravir//emtricitabine/tenofovir (B/F/TAF; antiretroviral treatment naïve, changing treatment, virological failure)

Exclusion Criteria:

* Pregnant women
* People living with HIV (PLHIV) living in institutionalization, with guardianship or impaired judgment (to avoid bias due to unability to assume responsibility for treatment compliance)
* PLHIV receiving assistance incompatible with the use of the electronic pillbox.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults living with HIV-1 receiving or starting once-daily B/F/TAF-based antiretroviral therapy
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with virological failure at 6 months | 6 months
  Virological failure is defined as a confirmed plasma viral load >50 copies/mL (HIV RNA)

SECONDARY OUTCOMES:
Proportion of patients with virological failure at 12 months | 12 months
  • Virological failure at 12 months as defined in Primary Outcome Measure
Proportion of patients with side-effect | 6-12 months
  • Side-effect rate measured by CTCAE V.5
Proportion of patients with emerging drug resistance mutations | 6-12 months
  • Emergence of drug resistance mutations according to ANRS AC11 in case of virological failure
Proportion of patients with good quality of life | 6-12 months
  • Quality of life measured by questionnaires (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent HOCQUELOUX, M.D., Principal Investigator — CHU d'Orléans (France); Jean-Jacques PARIENTI, M.D., PhD, Study Director — CHU de Caen (France)
Locations (8):
- France (8):
  - CHU de Caen, Caen
  - CHD Vendée, La Roche-sur-Yon
  - Hôpitaux Civils de Lyon, Lyon
  - CHU de Nantes, Nantes
  - CH de Niort, Niort
  - CHU d'Orléans, Orléans
  - CHU Pitié-Salpétrière, Paris
  - CHU de Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing may be discussed on a case-by-case basis and will be decided by the BICTECAPS scientific committee